CLINICAL TRIAL: NCT02654834
Title: Oxidative Stress Status During Anesthesia in Pediatric Surgical Room Staff Versus Non-operating Room Personnel: Pilot Study
Brief Title: Oxidative Stress in OR Personnel
Status: Withdrawn | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Haleh Saadat, Director of Complementary and Alternative Medicine, Nationwide Children's Hospital
Other Study IDs: IRB14-00098
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Oxidative Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two 5 mL blood samples collected at the start of a work week and at the end of a work week.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pediatric Operating Room (OR) Staff: OR Staff exposed to nitrous oxide, and other volatile anesthetics
  Interventions: Other: Exposure to nitrous oxide or other volatile anesthetics
- Pediatric Intensive Care Unit (ICU) Staff: ICU Staff unexposed to any volatile anesthetics

INTERVENTIONS:
Other: Exposure to nitrous oxide or other volatile anesthetics — No intervention, but routine work-place exposure to volatile anesthetics
  Groups: Pediatric Operating Room (OR) Staff

SUMMARY:
The purpose of this study is investigate to the effect(s) of chronic occupational exposure to N20 and volatile anesthetics on the extent of oxidative stress (DNA damage and the generation of the biochemical markers) in operating room staff, with different levels of exposure to halogenated hydrocarbons, in comparison to unexposed controls (Intensive Care Staff), and to determine the relationship between the degree of oxidative stress and psychological stress, as assessed by validated psychometric measures.

DETAILED DESCRIPTION:
This is a single blinded randomized, controlled and prospective clinical trial comparing oxidative stress status in two groups.

Subjects in two groups will be matched for gender, age, smoking habit and employment duration and will be randomized into one of the two groups of:

1. Pediatric OR Staff, and
2. control (e.g; ICU staff)

Biomarkers of oxidative stress will be measured in two different time points in each subject, (Monday Morning and, Friday afternoon of that same week->40 hours in Operating room or Intensive Care Unit).

The relationship between oxidative stress and psychological stress will also be assessed by validated psychometric measures.

ELIGIBILITY:
Inclusion Criteria:

1. CHOR-Staff who work > 40 hours per week in the operating rooms (Anesthesiologists, CRNA, Surgeons, Nurses)
2. NOR- Intensive Care Unit Staff who work > 40 hours per week in Intensive care unit (Physicians, Nurses, APN'S)

Exclusion Criteria:

Staff with the following history will be excluded:

1. Therapeutic exposure to radiation
2. On chemotherapeutic agents
3. History of General Anesthesia during the past two years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Twenty operating room staff and twenty intensive care unit staff (40 Total Participants)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Oxidative Stress | During exposure to volatile anesthetics over the course of a week in the work-place
  The extent of oxidative stress (DNA damage and the generation of the biochemical markers) in operating room staff with different levels of exposure to halogenated hydrocarbons, in comparison to unexposed controls.

SECONDARY OUTCOMES:
Psychological Stress | During exposure to volatile anesthetics over the course of a week in the work-place
  To determine the relationship between oxidative stress and psychological stress, as assessed by validated psychometric measures.

CONTACTS AND LOCATIONS:
Overall Officials: Haleh Saadat, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No